CLINICAL TRIAL: NCT03713866
Title: Peri-Procedural Transmural Electrophysiological Imaging of Scar-Related Ventricular Tachycardia
Brief Title: Peri-Procedural Transmural Electrophysiological (EP) Imaging of Scar-Related Ventricular Tachycardia
Acronym: ECGI-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Sapp (Other)
Collaborators: Nova Scotia Health Authority (Other); Rochester Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, John Sapp, Staff Cardiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAPP006
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Ventricular Tachycardia; Myocardial Infarction
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EP Imaging and Testing (Experimental): MRI images,120 lead body surface mapping and NIPS testing will be completed to correlate areas of VT scar.
  Interventions: Diagnostic Test: EP Imaging and Testing

INTERVENTIONS:
Diagnostic Test: EP Imaging and Testing — Magnetic Resonance Imaging: pre-procedure imaging is standard care prior to catheter ablation procedures for VT to document anatomy of the heart.
  120-Lead Body Surface Mapping: a 120-lead ECG will be recorded using a standardized mapping protocol. 120 disposable radiolucent silver chloride (Ag/AgCl) surface electrodes will be placed on the torso in 18 strips and connected via cables to an advanced acquisition system.
  Noninvasive programmed stimulation (NIPS) study will be performed using the patient's implanted defibrillator, and is part of standard practice during a VT catheter ablation.

SUMMARY:
Ventricular tachycardia (VT) contributes to over 350,000 sudden deaths each year in the US. Malignant VTs involve an electrical "short circuit" in the heart, formed by narrow channels of surviving tissue inside myocardial scar. An important treatment is to use catheter ablation to "block" the channel that forms the circuit. Effective ablation requires imaging guidance to visualize the VT circuit relative to scar structures in 3D. Unfortunately, with conventional catheter mapping, up to 90% of the VT circuits are too short-lived to be mapped. For the 10% "mappable" VTs, their data are only available during ablation and limited to one ventricular surface. This inadequacy of functional VT data largely limits the knowledge about scar-related VT and ablation strategies, and reduces the ability of clinicians to identify ablation targets and assess ablation outcome.

The central hypothesis of this proposal is that functional VT data, integrated with CT or MRI scar data in 3D, can improve VT ablation efficacy with pre-procedural identification of ablation targets and post-procedural mechanistic elucidation of ablation failure. This research builds on the rapidly increasing clinical interest in electrocardiographic imaging (ECGi), an emerging technique that obtains cardiac electrical activity through inverse reconstructions from ECGs. The specific objective is to push the boundary of ECGi to provide - as a conjunction to intra-procedural catheter mapping - pre-ablation and post-ablation imaging of functional VT circuits integrated with 3D scar structure.

DETAILED DESCRIPTION:
Electrocardiographic imaging (ECGi) is an emerging technique to image cardiac electrical activity through inverse reconstructions from body-surface ECGs. After 40 years of active research, the potential of ECGi as a noninvasive adjunct to catheter mapping is gaining rapid attention in the clinical community.

A total of 40 consecutive post-infarction VT patients will be prospectively enrolled and recruited from those who have been referred for catheter ablation of scar-related VT. Within 7 days before the ablation procedure, these patients will undergo noninvasive cardiac CT or MRI imaging and noninvasive programmed stimulation (NIPS) study with simultaneous 120-lead body- surface ECG mapping (pre-ablation NIPS). MRI will be performed for patients with implantable defibrillators for whom it is considered safe to do so. CT imaging will be performed for those with Implantable Cardioverter Defibrillators (ICDs) which are not MRI compatible.

At the time of scheduled ablation, all patients will undergo standard catheter mapping and ablation procedure as a part of standard care. Within 7 days after the ablation procedure, the patients will undergo cardiac MRI imaging and noninvasive programmed stimulation (NIPS) with simultaneous 120-lead body-surface ECG mapping (post-ablation NIPS). For patients who cannot undergo MRI, CT imaging will not be repeated.

At 6 months after the procedure, a follow-up will occur as a part of standard care where outcome data regarding the chronic success of the ablation procedure will be collected and ICD interrogation will be performed. No imaging or mapping is planned at the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* One or more episodes of sustained monomorphic VT
* Referred for catheter ablation
* Previously implanted ICD
* Signed the patient informed consent form
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Have estimated Glomerular Filtration Ratio (eGFR) less than 30
* Have a life expectancy less than 6 months or are listed for heart transplantation at time of inclusion
* Are pregnant
* Are on IV inotropic agents
* Have any contraindication to catheter ablation (including but not limited to mechanical prosthetic aortic and mitral valves, known protruding Left Ventricular (LV) thrombus
* New York Heart Association (NYHA) functional class IV
* Had ST wave elevation myocardial infarction within < 1 month
* Unwilling or unable to undergo cardiac MRI scan AND unwilling or unable to undergo cardiac CT scan (e.g. contrast allergy).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Termination of Ventricular Tachycardia | Less than 10 minutes post ablation
  The heart rhythm will be monitored continually with ECG electrodes to ascertain whether VT terminates with ablation.
VT recurrence rate | Less than 6 months post procedure
  Any recurring VT occurring within 6 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: John L Sapp, MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QEII HSC, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No